CLINICAL TRIAL: NCT02595892
Title: Phase 2 Study of M6620 (VX-970) in Combination With Gemcitabine Versus Gemcitabine Alone in Subjects With Platinum-Resistant Recurrent Ovarian or Primary Peritoneal Fallopian Tube Cancer
Brief Title: Gemcitabine Hydrochloride Alone or With M6620 in Treating Patients With Recurrent Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01910; NCI-2015-01910 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-724; 9944 (Other: Dana-Farber - Harvard Cancer Center LAO); 9944 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Serous Tumor; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — berzosertib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (gemcitabine hydrochloride) (Active Comparator): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover to Arm II.
  Interventions: Drug: Gemcitabine; Drug: Gemcitabine Hydrochloride
- Arm II (gemcitabine, ATR kinase inhibitor M6620) (Experimental): Patients receive gemcitabine hydrochloride as in Arm I and ATR kinase inhibitor M6620 IV over 60-90 minutes on days 2 and 9. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Berzosertib; Drug: Gemcitabine; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
  Arms: Arm II (gemcitabine, ATR kinase inhibitor M6620)
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011

SUMMARY:
This randomized phase II trial studies how well ATR kinase inhibitor M6620 (M6620) and gemcitabine hydrochloride work compared to standard treatment with gemcitabine hydrochloride alone in treating patients with ovarian, primary peritoneal, or fallopian tube cancer that has come back after a period of improvement (recurrent). ATR kinase inhibitor M6620 may stop the growth of tumor cells by blocking an enzyme needed for cell growth, and may also help gemcitabine hydrochloride work better. Gemcitabine hydrochloride is a drug used in chemotherapy that works to stop the growth of tumor cells by blocking cells from growing and repairing themselves, causing them to die. It is not yet known whether adding ATR kinase inhibitor M6620 to standard treatment with gemcitabine hydrochloride is more effective than gemcitabine hydrochloride alone in treating patients with ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess and compare progression free survival (PFS) between gemcitabine (gemcitabine hydrochloride)/M6620 (VX-970) and gemcitabine alone arms.

SECONDARY OBJECTIVES:

I. Determine and compare overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) between gemcitabine/M6620 (VX-970) and gemcitabine alone arms.

II. Determine and compare the safety profile of gemcitabine/M6620 (VX-970) and gemcitabine alone regimens.

III. Assess and compare PFS at 6 months between gemcitabine/M6620 (VX-970) and gemcitabine alone arms.

IV. Determine and compare the clinical benefit rate (CBR) between gemcitabine/M6620 (VX-970) and gemcitabine alone arms.

V. Determine and compare the duration of response (DOR) between gemcitabine/M6620 (VX-970) and gemcitabine alone arms.

VI. Determine and compare cancer antigen (CA)125 reduction by >= 50% between gemcitabine/M6620 (VX-970) and gemcitabine alone arms.

VII. Determine and compare overall survival (OS) between gemcitabine/M6620 (VX-970) and gemcitabine alone arms.

VIII. Determine the ORR for subjects in the gemcitabine alone arm who cross over to the gemcitabine/M6620 (VX-970) arm.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover to Arm II.

ARM II: Patients receive gemcitabine hydrochloride as in Arm I and ATR kinase inhibitor M6620 IV over 60-90 minutes on days 2 and 9. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed high grade serous ovarian or primary peritoneal or fallopian tube cancer; platinum resistant disease is defined as progression within 6 months after last platinum regimen
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam; measurable disease by RECIST version (v)1.1 with at least one measurable target lesion
* Prior therapy: No line limit but no more than 1 prior regimens in the platinum resistant setting; no prior treatment targeting the ATR/checkpoint kinase 1 (CHK1) pathway and no prior gemcitabine as single agent; hormonal therapies immunotherapy, and antiangiogenic therapies (as single agents) do not count as lines; poly (adenosine diphosphate [ADP]-ribose) polymerases (PARP)-inhibitors count as a line of therapy unless given in the maintenance setting; PARP-inhibitors given as maintenance after platinum therapy do not count as a line of therapy; prior carboplatin/gemcitabine is allowed provided that there was no disease progression within 12 months after completion of the carboplatin/gemcitabine regimen; subjects may begin protocol treatment at least 4 weeks or 5 half-lives, whichever is shorter, after their last dose of chemotherapy or hormonal therapy, assuming they are otherwise eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky >= 70%)
* Life expectancy of greater than 6 months
* Leukocytes >= 3,000/mcL (within 2 weeks prior to initiation of study treatment)
* Absolute neutrophil count >= 1,500/mcL (within 2 weeks prior to initiation of study treatment)
* Platelets >= 100,000/mcL (within 2 weeks prior to initiation of study treatment)
* Total bilirubin within normal institutional limits (within 2 weeks prior to initiation of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (within 2 weeks prior to initiation of study treatment)
* Creatinine =< upper limit of institutional normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (within 2 weeks prior to initiation of study treatment)
* Confirmation of availability of a formalin-fixed, paraffin-embedded (FFPE) tumor specimen with adequate tumor tissue (either one paraffin embedded tissue block OR 10 5-micron unstained slides from the block on regular [non-plus] slides and 1 hematoxylin and eosin [H&E] slide)
* All acute, clinically significant treatment-related toxicity from prior therapy, except for alopecia, must have resolved to grade =< 1 prior to study entry
* At least 4 weeks since major surgery or radiation therapy
* The effects of M6620 (VX-970) on the developing human fetus are unknown; for this reason and because deoxyribonucleic acid (DNA) damage inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 6 months after completion of study; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* No known hypersensitivity or contraindication to the components of study treatment (M6620 [VX-970], gemcitabine)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with primary platinum refractory disease, defined as progression while first line platinum based chemotherapy
* Patients who have had chemotherapy within 4 weeks or five half-lives, whichever is shorter, (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have had radiotherapy within 4 weeks
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; a scan to confirm the absence of brain metastasis is not required
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 (VX-970) or gemcitabine
* M6620 (VX-970) is primarily metabolized by CYP3A4; therefore concomitant administration with strong inhibitors or inducers of CYP3A4 should be avoided; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of; patients receiving any medications or substances that are inhibitors or inducers of cytochrome P450 3A (CYP3A4 enzyme) are ineligible; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because M6620 (VX-970) and/or gemcitabine are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620 (VX-970) and/or gemcitabine, breastfeeding should be discontinued if the mother is treated with M6620 (VX-970) and/or gemcitabine
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with M6620 (VX-970) and/or gemcitabine; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2026-08-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis A Konstantinopoulos, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (17):
- United States (17):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

REFERENCES:
- [Derived] Konstantinopoulos PA, Cheng SC, Wahner Hendrickson AE, Penson RT, Schumer ST, Doyle LA, Lee EK, Kohn EC, Duska LR, Crispens MA, Olawaiye AB, Winer IS, Barroilhet LM, Fu S, McHale MT, Schilder RJ, Farkkila A, Chowdhury D, Curtis J, Quinn RS, Bowes B, D'Andrea AD, Shapiro GI, Matulonis UA. Berzosertib plus gemcitabine versus gemcitabine alone in platinum-resistant high-grade serous ovarian cancer: a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2020 Jul;21(7):957-968. doi: 10.1016/S1470-2045(20)30180-7. Epub 2020 Jun 15. PMID 32553118

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Started | 36 | 34
Number of Participants From Arm I Who Crossed-over to Arm II | 15 | 0 (Not applicable since Arm II patients were not able to cross-over to Arm I.)
Completed | 36 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620) | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Median (Full Range); unit: Years] | 68.1 [46.8 to 75.2] | 60.9 [50.2 to 76.3] | 63.7 [46.8 to 76.3]
Sex: Female, Male [Count of Participants; unit: Participants] — Only females were eligible for participation given the disease being studied.
  Participants
    Female | 36 | 34 | 70
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 34 | 30 | 64
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 30 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
The Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status Scale was used to clinically grade participants at baseline. The protocol required participants to have an ECOG of 0 or 1 to be eligible for the study. The following language of Grades 0 and 1 were used by investigators when assessing participants:"0 Normal activity: Fully active, able to carry on all pre-disease performance without restriction" and "1 Symptoms, but ambulatory: Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work)."
  Participants
    0 | 22 | 20 | 42
    1 | 14 | 14 | 28
Stage at Diagnosis [Count of Participants; unit: Participants] — Staging was based on the FIGO (International Federation of Gynecology and Obstetrics) system where higher stagers are associated with worse outcomes.
  Participants
    II | 0 | 2 | 2
    III | 16 | 18 | 34
    IV | 14 | 9 | 23
    Unknown | 6 | 5 | 11
Previous Therapy Lines [Count of Participants; unit: Participants]
  1 | 10 | 3 | 13
  2 | 18 | 20 | 38
  3 | 5 | 6 | 11
  4 | 2 | 4 | 6
  5 | 0 | 1 | 1
  8 | 1 | 0 | 1
Previous Therapy Lines in Platinum Resistant Setting [Count of Participants; unit: Participants]
  1 | 11 | 14 | 25
  0 | 25 | 20 | 45
Previous Poly Adenosine Diphosphate-Ribose Polymerase (PARP) Inhibitor [Count of Participants; unit: Participants]
  Yes | 7 | 11 | 18
  No | 29 | 23 | 52

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was summarized using Kaplan-Meier analyses and compared between the two arms using the logrank test. Additionally, PFS was analyzed using a Cox Proportional Hazards Model, including the stratification factor, and will be used to estimate the hazard ratio of the gemcitabine hydrochloride (gemcitabine)/ataxia telangiectasia mutated and Rad3-related (ATR) kinase inhibitor M6620 (formerly VX-970) arm relative to the gemcitabine alone arm and the associated 90% confidence interval. Disease progression, per protocol, is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the diameters of target lesions, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Number of days from the day the subject received the first dose of protocol therapy to the date of documented progressive disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or death (regardless of cause), assessed up to 3 years
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 36 | 34
Weeks | 14.7 [9.7 to 36.7] | 22.9 [17.9 to 72.0]
Statistical Analysis 1: Comparison: Arm I (Gemcitabine Hydrochloride) vs Arm II (Gemcitabine, ATR Kinase Inhibitor M6620); Test type: Other; p = 0.044, Log Rank; Hazard Ratio (HR) = 0.57, 90% CI 2-sided [.33 to .98]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Defined as the percentage of subjects achieving a response rating of complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors (RECIST) in the whole population. Per RECIST v1.1 definitions for target lesions and assessed by conventional CT and MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the diameters of target lesions; Overall Response (OR) = CR + PR. ORR was summarized by counts (percentages) in each Arm.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 36 | 34
Participants | 4 | 1

3. Secondary Outcome: Progression Free Survival at 6 Months (PFS-6)
Description: Assessed and compared PFS-6 between gemcitabine/VX-970 and gemcitabine alone arms
Time Frame: Number of days from the day the subject received the first dose of protocol therapy to the date of documented progressive disease by RECIST version 1.1 or death (regardless of cause), assessed at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 36 | 34
Participants | 13 | 17

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of subjects achieving a response rating of stable disease >= 4 months, partial response (PR), or complete response (CR). Subject demographic and baseline characteristics will be summarized by mean, standard deviation, median, minimum, and maximum for continuous variables; and by counts and percentages for categorical variables. Summaries will be provided separately for each treatment group. Treatment group comparisons in CBR will be evaluated using logistic regression and expressed as odds ratios with associated 90% confidence intervals. In the event that rates are low, comparisons will be based on Fisher's exact test.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 36 | 34
Participants | 9 | 12
Statistical Analysis 1: Comparison: Arm I (Gemcitabine Hydrochloride) vs Arm II (Gemcitabine, ATR Kinase Inhibitor M6620); Test type: Other; p = 0.44, Fisher Exact; Two-Sided Fisher's exact test

5. Secondary Outcome: Objective Response Rate by Platinum Free Status
Description: Objective response rate by platinum-free status includes only informational summaries (counts of participants who met the categories outlined below) without formal statistical comparisons.
Time Frame: Up to 3 years
Population: The rows in the data table below represent the patients within the specified platinum-free interval category who experienced an objective response.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 36 | 34
Participants
  Patients who experienced an ORR with a platinum-free interval ≤3 months: number analyzed (Participants) | 13 | 13
  Patients who experienced an ORR with a platinum-free interval ≤3 months | 1 | 1
  Patients who experienced an ORR with a platinum-free interval 3-6 months: number analyzed (Participants) | 23 | 21
  Patients who experienced an ORR with a platinum-free interval 3-6 months | 3 | 0

6. Secondary Outcome: Percentage of Patients With a Reduction in CA-125
Description: Determined and compared CA125 reduction by > 50% between gemcitabine/VX-970 and gemcitabine alone arms.
Time Frame: CA-125 serum samples were collected from participants in both Arms I and II at baseline, on Day 1 of each cycle, and at the end-of-study treatment visit, assessed up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 36 | 34
Participants | 9 | 9

7. Secondary Outcome: Overall Survival (OS)
Description: Assessed and compared OS between gemcitabine/VX-970 and gemcitabine alone arms.
Time Frame: Number of weeks from the date of registration until date of death (regardless of cause), assessed up to 3 years.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 36 | 34
Weeks | 43.0 [34.4 to 67.9] | 59.4 [33.7 to 86.6]

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Determined and compared the safety profile of gemcitabine/VX-970 and gemcitabine alone regimens.
Time Frame: AE checks occurred on D1 and D8 of each cycle for up to 2 years and at the Final Treatment Visit. Patients who were removed from study treatment for unacceptable AEs were followed until resolution/stabilization of the AE up to 3 years, or until death.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 36 | 34
Participants | 10 | 9

9. Secondary Outcome: Duration of Response
Description: Duration of response was evaluated at the first instance of CR or PR through the earliest assessment of progressive disease, death, or the last follow-up where the subject had not yet progressed from her prior response. Informational summaries without formal statistical comparisons were produced.
Time Frame: Assessed for up to 3 years.
Population: Duration of response was evaluated only for patients who showed a CR or PR. Subjects who had a best response of SD, progressive disease, or were removed from treatment before the first assessment of response were not evaluated for duration of response.
Measure: Number; unit: Weeks
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)
Number analyzed (Participants) | 4 | 1
Weeks
  Patient 1: number analyzed (Participants) | 1 | 0
  Patient 1 | 10 |
  Patient 2: number analyzed (Participants) | 1 | 0
  Patient 2 | 6 |
  Patient 3: number analyzed (Participants) | 1 | 0
  Patient 3 | 18 |
  Patient 4: number analyzed (Participants) | 1 | 0
  Patient 4 | 27 |
  Patient 5: number analyzed (Participants) | 0 | 1
  Patient 5 |  | 7

ADVERSE EVENTS:
Time Frame: AE checks occurred on D1 and D8 of each cycle for up to 2 years and at the Final Treatment Visit. Patients who were removed from study treatment for unacceptable AEs were followed until resolution/stabilization of the AE up to 3 years, or until death.
Description: Safety and adverse events were assessed on day 1 and day 8 of each cycle and were graded according to the NCI Common Terminology Criteria for Adverse Events version 4.0.
Groups:
- Arm II (Gemcitabine, ATR Kinase Inhibitor M6620) After Crossover: Per protocol, participants could cross-over from "Arm I (Gemcitabine Hydrochloride)" to "Arm II (Gemcitabine, ATR Kinase Inhibitor M6620)" if disease progression was experienced. This adverse event arm demonstrates the events which occurred during Arm II treatment for the 15 total participants who crossed over.
Arm/Group | Arm I (Gemcitabine Hydrochloride) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620) After Crossover
All-Cause Mortality (participants affected / at risk) | 18/36 | 24/34 | 11/15
Serious Adverse Events (participants affected / at risk) | 10/36 | 9/34 | 3/15
Other Adverse Events (participants affected / at risk) | 36/36 | 34/34 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Gemcitabine Hydrochloride) (N=36) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620) (N=34) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620) After Crossover (N=15)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Platelet count decrease (Investigations) | 1 | 4 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Addisonian crisis (Endocrine disorders) | 0 | 1 | 0
Neutrophil count decrease (Blood and lymphatic system disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Gemcitabine Hydrochloride) (N=36) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620) (N=34) | Arm II (Gemcitabine, ATR Kinase Inhibitor M6620) After Crossover (N=15)
Anemia (Blood and lymphatic system disorders) | 24 | 22 | 7
Blood Bilirubin Decreased (Blood and lymphatic system disorders) | 1 | 0 | 0
Decreased BUN (Blood and lymphatic system disorders) | 0 | 1 | 0
Decreased Hematocrit (Blood and lymphatic system disorders) | 2 | 2 | 1
Decreased MCHC (Blood and lymphatic system disorders) | 2 | 0 | 0
Decreased RBC (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Increased Absolute Immature Granulocyte (Blood and lymphatic system disorders) | 0 | 1 | 0
Increased MCV (Blood and lymphatic system disorders) | 1 | 0 | 0
Increased RDW (Blood and lymphatic system disorders) | 1 | 1 | 0
Increased Red Blood Cell Distribution (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 6 | 1 | 2
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 21 | 23 | 4
Platelet Count Decreased (Blood and lymphatic system disorders) | 5 | 13 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
White Blood Cell Decreased (Blood and lymphatic system disorders) | 8 | 8 | 2
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Increased BUN (Endocrine disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 6 | 1
Decreased Appetite (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 8 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis Oral (Gastrointestinal disorders) | 1 | 6 | 1
Nausea (Gastrointestinal disorders) | 17 | 19 | 6
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Mucositis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 11 | 4
Chills (General disorders) | 2 | 5 | 1
Edema Limbs (General disorders) | 7 | 1 | 0
Fatigue (General disorders) | 21 | 22 | 4
Fever (General disorders) | 2 | 7 | 2
Flu Like Symptoms (General disorders) | 4 | 4 | 0
Infusion Related Reaction (General disorders) | 1 | 2 | 0
Infusion Site Extravasation (General disorders) | 0 | 2 | 0
Injection Site Reaction (General disorders) | 0 | 1 | 0
Localized Edema (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 1 | 0
Allergic Reaction (Immune system disorders) | 0 | 1 | 0
Mucosal Infection (Infections and infestations) | 1 | 0 | 0
Rash Pustular (Infections and infestations) | 0 | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 3 | 0
Alanine Aminotransferase Increased (Investigations) | 7 | 10 | 2
Alkaline Phosphatase Increased (Investigations) | 1 | 1 | 3
Aspartate Aminotransferase Increased (Investigations) | 8 | 12 | 2
Cardiac Troponin T Increased (Investigations) | 1 | 0 | 0
Creatinine Increased (Investigations) | 1 | 1 | 1
Lipase Increased (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 7 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Leg Cramping (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0
Restless Legs (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 8 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1 | 0
Unbalanced (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 5 | 1
Derm Other-left Wrist (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Itch (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nonfluid Filled Blisters On Thumbs (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 4 | 0
Red Painful Finger/thumbs (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Red Painful Thumbs And Toes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Thromboembolic Event (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT02595892/Prot_SAP_000.pdf